CLINICAL TRIAL: NCT05413239
Title: Improving Glycemia & Reducing Diabetes Distress in Adolescents & Young Adults With T1D: Healthy And Positive Pathways for Young People With Type 1 Diabetes (HAPPY T1D)
Brief Title: Healthy And Positive Pathways for Young People With Type 1 Diabetes (HAPPY T1D)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Stanford University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00000154; R01DK129479 (NIH)
Record Dates: First submitted 2022-06-07; First posted 2022-06-09 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The Intervention Group will receive the monthly intervention sessions during the first year of the study.
  Interventions: Behavioral: Psychoeducation to reduce diabetes distress and improve glycemic outcomes
- Control Group (No Intervention): The Control Group will receive the monthly intervention sessions during the second year of the study (after assessment of primary outcomes at 1 year).

INTERVENTIONS:
Behavioral: Psychoeducation to reduce diabetes distress and improve glycemic outcomes — The intervention includes two types of sessions - those targeting an improvement in glycemic outcomes and those targeting a reduction in diabetes distress. Evidence indicates that psychoeducation and support are needed to improve self-care behaviors and optimize use of advanced diabetes technologies, which, in turn, can help improve diabetes control while also reducing diabetes distress. Participants will receive 4 one-on-one glycemic sessions and 8 one-on-one distress sessions, each lasting ~30 minutes. Sessions will be conducted in-person or remotely. The virtual sessions are intended to provide the extra psychoeducation and support needed for this high risk group without increasing the burden associated with frequent face-to-face sessions.
  Arms: Intervention Group

SUMMARY:
In this 2-year randomized clinical trial, we will implement and assess the impact of a behavioral/psychoeducational intervention to reduce diabetes distress and improve glycemic outcomes in adolescents and young adults, aged 14-25 years, with T1D in order to optimize their short-term and long-term health.

DETAILED DESCRIPTION:
In this study, we will recruit 180 adolescents and young adults (ages 14-25) with type 1 diabetes for at least 1 year and suboptimal diabetes control (A1c 7-13%) to participate in a 2-year randomized clinical trial aimed at reducing diabetes distress and improving glycemic outcomes. Adolescents and young adults with type 1 diabetes represent a population that often has uncontrolled diabetes with elevated A1c levels and experiences diabetes distress, making such patients ideal for this study. Participants will be randomly assigned to one of two groups (control or intervention). The intervention group will participate in monthly intervention sessions with a research assistant during the first year of the study. Four sessions will focus on improving glycemic outcomes and 8 sessions will focus on reducing diabetes distress. The sessions will be conducted face-to-face or remotely. To ensure adequate recruitment and retention, the control group will participate in the intervention sessions during the second year of the study. Participants in both groups will use continuous glucose monitoring (CGM), with CGM data downloaded every 3 months. Participants in both groups will complete surveys and have A1c measured every 6 months. We will compare the two groups on percent time in target glucose range (70-180 mg/dL), A1c, and diabetes distress from baseline to 1 year. We hypothesize that the intervention group will have an improvement in percent time in range, A1c, and diabetes distress, compared with the control group.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-25 years
* Diagnosis of type 1 diabetes (according to ADA criteria)
* Type 1 diabetes duration ≥12 months
* A1c 7-13%
* Smartphone or regular access to wifi via computer
* Fluency in English at a 5th grade level or higher (based on investigator assessment of grade level in school or highest grade level achieved and presence in mainstream academic classes)

Exclusion Criteria:

* Physical or mental health condition that in the determination of the investigators may limit the ability to fully participate in the study (e.g., autism)
* Participation in another intervention study within the last 3 months
* Currently pregnant or intending to become pregnant during the study (assessed by self-report)

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 191 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Time in Range (TIR) | 0, 3, 6, 9, 12, 15, 18, 21, and 24 months
  CGM data will be downloaded every 3 months to assess percent time in range (TIR) (70-180 mg/dL). The primary outcome will be change in TIR from 0 to 12 months for intervention group vs. control group.

SECONDARY OUTCOMES:
A1c | 0, 6, 12, 18, and 24 months
  A1c will be assessed every 6 months. Blood samples will be collected locally using uniform procedures and sent to the central laboratory at the University of Minnesota for analysis. Change in A1c from 0 to 12 months will be compared within and between the intervention group and control group.
Diabetes distress | 0, 6, 12, 18, and 24 months
  Diabetes distress will be assessed every 6 months using the validated Problem Areas in Diabetes - Pediatric survey (PAID-Peds) and the Diabetes Distress Scale. Change in diabetes distress from 0 to 12 months will be compared within and between the intervention group and control group.
Attitudes toward diabetes device use | 0, 6, 12, 18, and 24 months
  Attitudes toward diabetes device use will be assessed every 6 months using the validated Glucose Monitoring Satisfaction Survey and the Diabetes Technology Attitudes Scale. Change in attitudes toward device use from 0 to 12 months will be compared within and between the intervention group and control group.

OTHER OUTCOMES:
Hypoglycemia experience | 0, 6, 12, 18, and 24 months
  Fear of hypoglycemia and confidence in hypoglycemia management will be assessed every 6 months with the Fear of Hypoglycemia Screener and the Hypoglycemia Confidence Scale. Change in hypoglycemia experience from 0 to 12 months will be compared within and between the intervention group and control group.
Health-related quality of life | 0, 6, 12, 18, and 24 months
  Health-related quality of life will be assessed every 6 months with the PROMIS Global Health Measure. Change in quality of life from 0 to 12 months will be compared within and between the intervention group and control group.
Diabetes incorporation/identity | 0, 6, 12, 18, and 24 months
  Diabetes incorporation/identity will be assessed every 6 months with the Accepting Diabetes And Personal Treatment (ADAPT) survey. Change in diabetes incorporation/identity from 0 to 12 months will be compared within and between the intervention group and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Lori M Laffel, MD, MPH, Principal Investigator — Joslin Diabetes Center; Korey K Hood, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - Joslin Diabetes Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
If we are able to remove all HIPAA-defined identifiers from the final data set to eliminate the possibility of deductive disclosure of participants with unusual characteristics, the investigators will make the final data set available to interested researchers according to the NIH Data Sharing Policy and the criteria below.
Time Frame: After all of the investigators' analyses, presentations, and publications of study findings are complete
Access Criteria: If it is determined that data can be shared, data will be made available upon request to qualified persons only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are complete.

DOCUMENTS (1):
  • Informed Consent Form (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/39/NCT05413239/ICF_000.pdf